CLINICAL TRIAL: NCT02424201
Title: Comparative Study on Effects of Sublingual Misoprostol in Addition to Standard Active Management of Third Stage of Labour in Low Risk Parturients in Lagos State University Teaching Hospital, Ikeja.
Brief Title: Comparative Study on the Effects of Sublingual Misoprostol in Addition to Standard AMTSL in Low Risk Parturients in LASUTH, Ikeja.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lagos State University (Other)
Responsible Party: Principal Investigator, Oyedeko Muyideen Oladipo, Doctor, Lagos State University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: LagosSU
Record Dates: First submitted 2015-04-18; First posted 2015-04-22 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Primary Postpartum Haemorrhage
Keywords: uterine atony
MeSH Terms: conditions — Uterine Inertia | interventions — Misoprostol; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study (Experimental): Intramuscular oxytocin 10 units, 400 micrograms of misoprostol
  Interventions: Drug: Misoprostol
- control (Other): Intramuscular oxytocin 10 units, 2 tablets of placebo which will be vitamin c
  Interventions: Drug: vitamin c

INTERVENTIONS:
Drug: Misoprostol — experimental
  Other Names: Cytotec
  Arms: study
Drug: vitamin c — control
  Other Names: ascorbic acid
  Arms: control

SUMMARY:
Postpartum haemorrhage is the leading cause of maternal haemorrhage globally. With active management of labour 3 to 16.5% of parturients still experience postpartum haemorrhage. Hence the need for an effective oxytocic in third stage of labour.

DETAILED DESCRIPTION:
This is a prospective randomized doubleblind controlled trial involving 660 consenting pregnant women. Eligible subjects will be ransomised into 2 groups of 330 participants. All patients will receive the standard oxytocin 10 units as part of the active management of third stage of labour. However, the study group will be administered sublingual 400 misoprostol while the control group will receive 2tablets of placebo (vitamin c). Measured mean blood loss will be comparee in the 2 groups using statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* singleton in longitudinal lie and cephalic presentation

Exclusion Criteria:

* refusal of consents, multiple gestation

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 660 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
mean blood loss | 1 hour of delivery

SECONDARY OUTCOMES:
number of participants with untowards effects | 1 hour of delivery

REFERENCES:
- [Derived] Ottun TA, Adewunmi AA, Rabiu AK, Olumodeji AM, Oladipo OM, Olalere HF. Misoprostol and oxytocin versus oxytocin alone in the active management of the third stage of labour: a randomised, double-blind, placebo-controlled trial. J Obstet Gynaecol. 2022 Jul;42(5):1048-1053. doi: 10.1080/01443615.2021.1995342. Epub 2021 Dec 27. PMID 34958620